CLINICAL TRIAL: NCT00892801
Title: A Phase I/II Study of RAD001 and Radiation Therapy in Patients With Brain Metastasis From Non-small Cell Lung Cancer (NSCLC)
Brief Title: Everolimus and Whole-Brain Radiation Therapy in Treating Patients With Brain Metastasis From Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to low accrual. Study was closed to accrual prematurely and did not continue on to Phase II.
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vicki Keedy, MD, Medical Director, Vanderbilt-Ingram Cancer Center, Clinical Trials Shared Resource; Assistant Professor, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0772; P30CA068485 (NIH); VU-VICC-THO-0772; IRB#090314
Record Dates: First submitted 2009-05-02; First posted 2009-05-05 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): RAD001 + radiation therapy
  Interventions: Drug: RAD001; Radiation: whole-brain radiation therapy

INTERVENTIONS:
Drug: RAD001 — Taken by mouth once a day, for 15 days, one day prior to initiation of whole brain radiation therapy at 5 or 10 mg/day during the phase I component. One of these doses will be selected as the maximum tolerable dose and will be selected for the phase II component
Radiation: whole-brain radiation therapy — Standard whole brain radiation therapy (WBRT) 30 Gy will be given in ten fractions.

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving everolimus together with whole-brain radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus and to see how well it works when given together with whole-brain radiation therapy in treating patients with brain metastasis from non-small cell lung cancer.

DETAILED DESCRIPTION:
Phase I is intended to determine the maximum tolerated dose. Study drug will be administered orally, once a day, for 15 days, one day prior to initiation of WBRT at 5 or 10 mg/day during the phase I component. One of these doses will be selected as the maximum tolerable dose and will be selected for the phase II component.

OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of everolimus when combined concurrently with whole-brain radiotherapy in patients with brain metastasis from stage IV non-small cell lung cancer. (Phase I)
* To evaluate the median survival of these patients treated with this regimen. (Phase II)

Secondary

* To assess the response rates in these patients. (Phase II)
* To assess the safety and tolerability of this regimen in these patients. (Phase II)
* To determine time to CNS (neurological) progression, confirmed by MRI, in these patients. (Phase II)
* To determine time to systemic (non-CNS) progression in these patients. (Phase II)

OUTLINE: This is a multicenter, dose-escalation study of everolimus.

Patients undergo 10 fractions of whole-brain radiotherapy (WBRT) beginning on day 0, 5 days per week, and receive oral everolimus once daily on days -1 to 13. Beginning 2 weeks after completion of WBRT, patients receive oral everolimus once daily for 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiographically confirmed brain metastases with histopathologically confirmed primary non-small cell lung cancer that will benefit from whole-brain radiotherapy
* Must have ≥ 1 measurable intracranial site of disease, according to RECIST criteria, that has not been previously treated with stereotactic radiation
* Must have stable extracranial disease for 4 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC > 1,500/mm³
* Platelets > 100,000/mm³
* Hemoglobin > 11 g
* BUN ≤ 25 mg
* Serum creatinine < 1.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 times ULN
* Serum transaminases ≤ 2 times ULN (< 5 times ULN if patient has liver metastases)
* Cholesterol ≤ 300 mg/dL
* Triglycerides ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No other malignancies within the past 3 years, except for adequately treated carcinoma in situ of the cervix or basal or squamous cell carcinomas of the skin
* No severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study, including any of the following:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within the past 6 months, or serious uncontrolled cardiac arrhythmia
  * Severely impaired lung function (i.e., FEV1 < 0.8 cc)
  * Uncontrolled diabetes as defined by fasting serum glucose ≥ 1.5 times ULN
  * Any active (acute or chronic) or uncontrolled infection/disorders
  * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
  * Liver disease, such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
* No known history of HIV seropositivity
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No active, bleeding diathesis
* No known hypersensitivity to everolimus or other rapamycin (i.e., sirolimus, temsirolimus) or to its excipients
* No history of noncompliance to medical regimens

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the acute toxicities of any prior therapy
* Prior surgical resection of a brain metastasis allowed

  * The extent of surgical resection in patients having prior resection of 1 of multiple metastases shall be documented as a biopsy, subtotal resection, or total resection as described by the operative report and/or post-operative imaging
* At least 3 weeks since prior major surgery or completion of extracranial radiation
* At least 3 weeks since prior and no concurrent systemic anticancer therapy, other than the study medications administered as part of this study protocol
* At least 6 weeks since prior nitrosoureas
* More than 1 week since prior and no concurrent immunization with attenuated live vaccines
* More than 3 weeks since prior chemotherapy
* No prior brain radiotherapy of any form
* No concurrent chronic treatment with systemic steroids or other immunosuppressive agents, except steroids for neurological stability following the diagnosis of brain metastases
* No prior treatment with an mTOR inhibitor
* No concurrent anti-vitamin K medication, except low dose coumarin
* No concurrent drugs or substances known to be inhibitors or inducers of the isoenzyme CYP3A
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 week DLT period
  Safety is measured by the rate of ≥ grade 3 hematological and non-hematologic study-related toxicities.
Median survival (phase II) | Off-study date.

SECONDARY OUTCOMES:
Intracranial response rate (phase II) | Off-treatment date.
Time to CNS (neurologic) progression (phase II) | Off-treatment date.
Time to systemic non-CNS progression (phase II) | Off-treatment date

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Keedy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee